CLINICAL TRIAL: NCT07360483
Title: Treatment of Hypertrophic Scars Using Fractional CO2 Laser Alone in Comparison With Adding Botulinum Toxin Either Through Intralesional Injection or Assisted Drug Delivery
Acronym: BTX and LADD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Fahim, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-257 2024
Record Dates: First submitted 2025-12-27; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hypertrophic Scars
Keywords: hypertrophic scar; LADD; botulinum toxin A
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Received Fractional CO2 Laser with Intralesional Botox injection (FL + Inj. Botox). (Active Comparator): * laser treatment was performed using ( DEKA SmartXide DOT, Italy). Treatment parameters included power (18-20W), dwell time (800-1000µs), spacing (500-600µm, 13% density), micro spot size (120µm), and 2-3 stacks, adjusted depending on scar height
  * For eye protection, eye goggles were used during the sessions. Patients were instructed to apply a full-spectrum sunscreen regularly. Topical antibiotic cream was applied twice per day for 5 days following the session, and emollients twice daily for two weeks
  * Immediately following laser treatment, Botulinum toxin type A (Botox Allergan, Irvine, CA; 100U vacuum-dried powder reconstituted in 2mL of sterile, preservative-free 0.9% saline to a concentration of 5U/0.1mL) was injected intralesionally into the scar tissue for Section 1.
    * A 24-gauge needle (0.3mm × 0.8mm) was used, and the injection was continued until slight blanching was visible. The dose was adjusted to 2.5 U/cm³ of the lesion, not exceeding 100 units per session
  Interventions: Drug: Botulinum toxin type A (Botox®, Allergan)
- Received Fractional CO2 Laser Only (FL Only). (Active Comparator): Fractional CO2 laser treatment was performed using ( DEKA SmartXide DOT, Italy). Treatment parameters included power (18-20W), dwell time (800-1000µs), spacing (500-600µm, 13% density), micro spot size (120µm), and 2-3 stacks, adjusted depending on scar height For eye protection, eye goggles were used during the sessions. Patients were instructed to apply a full-spectrum sunscreen regularly. Topical antibiotic cream was applied twice per day for 5 days following the session, and emollients twice daily for two weeks
  Interventions: Drug: Botulinum toxin type A (Botox®, Allergan)
- Received Fractional CO2 Laser with Botulinum Toxin Assisted Drug Delivery (topical) (FL + Topical Bo (Active Comparator): * Fractional CO2 laser treatment was performed using ( DEKA SmartXide DOT, Italy). Treatment parameters included power (18-20W), dwell time (800-1000µs), spacing (500-600µm, 13% density), micro spot size (120µm), and 2-3 stacks, adjusted depending on scar height (Tawfic et al., 2022). For eye protection, eye goggles were used during the sessions. Patients were instructed to apply a full-spectrum sunscreen regularly. Topical antibiotic cream was applied twice per day for 5 days following the session, and emollients twice daily for two weeks.
  * Immediately following laser treatment, Botulinum toxin type A (Botox Allergan, Irvine, CA; 100U vacuum-dried powder reconstituted in 2mL of sterile, preservative-free 0.9% saline to a concentration of 5U/0.1mL) -• Immediately following laser treatment for Section 3, topical Botulinum toxin (prepared at the same concentration 2.5 U/cm³ of the lesion as for intralesional injection and adjusted to 2.5 U/cm³) was applied to the treated area topically
  Interventions: Drug: Botulinum toxin type A (Botox®, Allergan)

INTERVENTIONS:
Drug: Botulinum toxin type A (Botox®, Allergan) — Fractional CO2 laser 10, 6000nm

SUMMARY:
The current study aimed to evaluate the effectiveness of fractional laser treatment alone and fractional laser combined with botulinum toxin A, delivered either through injections or topical application fractional laser-assisted drug delivery (FLADD) in hypertrophic burn scar

DETAILED DESCRIPTION:
Burn injuries represent a major global health concern, often resulting in long term physical, psychological, and social consequences. Among the most challenging sequelae are hypertrophic scars, which arise from abnormal wound healing characterized by fibroblast hyperactivity, excessive collagen deposition and impaired extracellular matrix remodeling. These scars not only compromise skin pliability and aesthetics but also restrict mobility, leading to functional disability and reduced quality of life.

Traditional management strategies including surgical excision, corticosteroid injections, silicone gel, pressure therapy, and radiation have shown variable efficacy, with high recurrence rates and limited patient satisfaction. In recent years, minimally invasive modalities such as fractional CO2 laser therapy have gained prominence for their ability to remodel scar tissue and improve texture. Concurrently, botulinum toxin type A (BTXA) has emerged as a promising antifibrotic agent, exerting its effects by reducing wound tension, modulating fibroblast activity, and regulating collagen synthesis.

The integration of fractional CO2 laser with BTXA, delivered either intralesionally or via laser assisted drug delivery, offers a novel therapeutic approach aimed at enhancing scar pliability, contour and patient comfort. This study investigates the comparative efficacy of these modalities in the treatment of post burn hypertrophic scars, providing evidence to guide optimized clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Scar Type: Clinically diagnosed hypertrophic burn scar not less than 4.5 cm
2. Minimum Scar Size: 4.5cm x 1 cm
3. Scar duration: At least 1 month old and not exceed 6 months.
4. Fitzpatrick Skin Type: II to IV
5. No Recent Scar Treatment: No scar treatment within the past 6 months
6. Healthy Skin: No active skin infections in the treatment area
7. Normal Neuromuscular Function: No history of neuromuscular disorders or medications affecting muscle function.

Exclusion Criteria:

* 1) Pregnancy /Lactation: Pregnant, lactating, or planning pregnancy within 6 months 2) patients did previous intervention for the scar for the last 6 months 3) Bleeding Disorders: Known cases of bleeding disorders 4) patients with allergic reaction to botulinum toxin or with neuromuscular junction diseases (eg, myasthenia gravis) 5) patients on medication that decrease neuromuscular transmission (eg, aminoglycosides, penicillamine, quinine, and calcium channel blockers).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Change in total Patient and Observer Scar Assessment Scale (POSAS) score for each scar section | Baseline and 3 months after the last treatment session
  The Patient and Observer Scar Assessment Scale (POSAS) include a 6-item Patient Scar Assessment Scale (score range 6-60) and a 5-item Observer Scar Assessment Scale (score range 5-50). Each item is scored from 1 (normal skin) to 10 (worst imaginable scar). Total scores are calculated by summing item scores. The primary endpoint is the change in POSAS total score (patient and observer components) from baseline to 3 months after the last treatment session for each of the three scar sections.
Change in Vancouver Scar Scale (VSS) total score | Baseline and 3 months after the last treatment session.
  The VSS evaluates four scar characteristics: pigmentation (0-2), vascularity (0-3), pliability (0-5), and height (0-3). Total VSS score ranges from 0 to 13, with higher scores indicating more severe scarring. The outcome is the change in total VSS score between baseline and 3 months after the final treatment session.

SECONDARY OUTCOMES:
Change in quantitative scar elevation measured by Antera 3D imaging | Baseline and 3 months after the last treatment session
  •Scar elevation (height above surrounding normal skin) will be measured in microns using the Antera 3D camera (Miravex, Dublin). The same region of interest (ROI) is analyzed at baseline and follow-up using the software's alignment/synchronization feature. The outcome is the change in mean elevation value (µm).
Change in scar roughness/texture measured by Antera 3D imagingChange in scar roughness/texture measured by Antera 3D imaging | Baseline and 3 months after the last treatment session.
  Surface texture irregularity will be quantified using Antera 3D software's roughness parameter, reported in microns. The same ROI is assessed at both visits to measure change in roughness.
Change in scar redness (oxyhemoglobin concentration) measured by Antera 3D imaging | Baseline and 3 months after the last treatment session.
  Antera 3D hemoglobin analysis quantifies vascularity using hemoglobin level and hemoglobin variation parameters. Results are expressed as numeric values representing vascularity intensity. The endpoint is the change in hemoglobin parameters from baseline.
Change in scar pigmentation (melanin concentration) measured by Antera 3D imaging | Baseline and 3 months after the last treatment session
  Melanin level and melanin variation are quantified through Antera 3D imaging. Numeric melanin values are compared between baseline and follow-up to determine improvement in hyperpigmentation.
Global Assessment Score (Independent Blinded Evaluator) | 3 months after the final treatment session
  A single blinded dermatologist will provide a global qualitative rating of scar improvement, integrating texture, vascularity, color, and height. Scores will be reported categorically using a 5-point scale:
  1. = No improvement,
  2. = Mild,
  3. = Moderate,
  4. = Marked,
  5. = Excellent improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Salah El-Mesidy, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Tawfik AA, Ali RA. Evaluation of botulinum toxin type A for treating post burn hypertrophic scars and keloid in children: An intra-patient randomized controlled study. J Cosmet Dermatol. 2023 Apr;22(4):1256-1260. doi: 10.1111/jocd.15634. Epub 2023 Jan 31. PMID 36718819
- [Background] Sabry, H.H., Hamed, A.M., & Ibrahim, E.A. (2020). Comparative Study between Intralesional and Topical Botulinum Toxin A Combined with Fractional Carbon Dioxide Laser in Treatment of Hypertrophic Scars and Keloids (Comparative study). Benha Journal of Applied Sciences, 5(3 part (2)), 187-189.